CLINICAL TRIAL: NCT04442698
Title: Tailored Bilio-Pancreatic Limb Length and Hemoglobin A1c Levels 10 Years Following Mini-Gastric Bypass Original Technique
Brief Title: Tailored Bilio-Pancreatic Limb and HbA1c 10 Years Post Mini-Gastric Bypass
Acronym: BPLLvHbA1c
Status: Completed | Type: Observational
Sponsor: Kular Hospital (Other)
Responsible Party: Principal Investigator, Dr. Robert Rutledge, Research Director, Kular Hospital
Other Study IDs: KularH
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Diabetes; Surgery
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic MGB post op patients: Diabetic MGB post op patients
  Interventions: Procedure: Mini-Gastric Bypass Original Technique

INTERVENTIONS:
Procedure: Mini-Gastric Bypass Original Technique — Follow up of the Surgical procedure outcomes in diabetics. Procedure Mini-Gastric Bypass Original Technique
  Other Names: One Anastomosis Bypass

SUMMARY:
Diabetes is now or soon will be a worldwide epidemic. Diabetes has impact on both healthcare costs in addition to the costs in human lives, suffering and disability. Treatment that lowers Hemoglobin A1c (HbA1c) improved outcomes. Studies have demonstrated that both general surgery and bariatric procedures may improve or reverse diabetes. In several studies the Billroth II reconstruction following gastrectomy was the most effective surgical technique in improving or reversing Diabetes. The purpose of this study is to analyze the outcomes of the Mini-Gastric Bypass-Original Technique (MGB-OT) version of the One Anastomosis Bypass (OAGB) to investigate the association of a "Tailored" Bilio-pancreatic Limb Length (BPLL) with the HbA1c changes.

DETAILED DESCRIPTION:
There is general agreement that Diabetes is now or soon will be a worldwide epidemic. Studies also make clear the devastating impact of diabetes on both healthcare costs in addition to the costs in human lives, suffering and disability. It is also clear that treatment that lowers Hemoglobin A1c (HbA1c) will result in improved outcomes proportional to the decrease, saving both lives and costs. Unfortunately medical and lifestyle therapy routinely result in less than ideal resolution of elevated HbA1c levels. Studies have demonstrated that both general surgery and bariatric procedures may improve or reverse diabetes. In several studies the Billroth II reconstruction following gastrectomy is the most effective surgical technique in improving or reversing Diabetes. The purpose of this study is to analyze the outcomes of the Mini-Gastric Bypass-Original Technique (MGB-OT) version of the One Anastomosis Bypass (OAGB) to investigate the association of a "Tailored" Bilio-pancreatic Limb Length (BPLL) with the HbA1c changes.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Gastric Bypass -Original Technique post operative patients

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having undergone Mini-Gastric Bypass -Original Technique post operative patients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c Levels (HbA1c) | 10 years
  HbA1c Levels
Delta Hemoglobin A1c Levels (HbA1c) | 10 years
  Delta HbA1c from Before to After MGB-OT surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kular Hospital, Khanna, Punjab, India

IPD SHARING:
Plan to Share IPD: No